CLINICAL TRIAL: NCT07359768
Title: SCAPIS 2 - Spectrum Study -CVD Risk Based on Microvascular Dysfunction
Brief Title: Non-invasive Microvascular Assessment in Individuals at High Risk of Cardiovascular Disease From the SCAPIS2 Study
Status: Recruiting | Type: Observational
Sponsor: HJN Sverige AB/Neko Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-01937-01; CIV-23-12-045355 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Microvascular Complications
Keywords: microvascular; non-invasive; microcirculation; spatial frequency domain imaging; cardiac magnetic resonance imaging; laser speckle contrast imaging; laser doppler flowmetry
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and serum samples. Approximately 25 ml of blood will be collected for analysis of various markers relevant to the study objectives, such as variables that may be associated with vascular function, inflammation, and metabolism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- O-CAD: O-CAD arm inclusion is based on burden of coronary atherosclerosis measure in computer tomography of coronary arteries (CCTA) as measured by coronary artery disease reporting and data system (CADRADS). If CAD-RADS is above or equal to 3, participant may be eligible for inclusion in O-CAD arm.
- ANOCA: ANOCA arm inclusion is dictated by presence of cardiac angina as defined by the rose questionnaire and CAD-RADS <3. Exclusion criteria are similar as to those for stress-CMR.
- Metabolic: Inclusion is dictated by prevalence of diabetes mellitus concomitantly present with metabolic syndrome with metabolic syndrome severity score higher than 4. Exclusion criteria are similar as to those for stress-CMR, alongside CAD RADS < 3 and no angina as defined by rose questionnaire.
- Left ventricular diastolic dysfunction: Inclusion is dictated by diastolic dysfunction as defined by British Society of Echocardiography. Exclusion criteria are similar as to those for stress- CMR, alongside CAD RADS < 3 and no angina as defined by rose questionnaire.

SUMMARY:
Microvascular dysfunction, particularly endothelial dysfunction, is increasingly recognized as a key mechanism underlying various cardiovascular diseases (CVD), including heart failure, ischemic heart disease, atherosclerosis, stroke, dementia, and kidney failure. Chronic low-grade inflammation linked to metabolic syndrome may further drive systemic microvascular impairment. Early detection of these subclinical processes using non-invasive assessments could facilitate timely interventions to prevent disease progression.

SCAPIS 2 Spectrum is a prospective observational sub-study of the Swedish Cardiopulmonary Bioimage Study (SCAPIS-2), recruiting approximately 900 subjects aged 60-75 years. The study is organized into five arms-obstructive coronary artery disease (O-CAD), angina with nonobstructive coronary arteries (ANOCA), metabolic syndrome with diabetes, left ventricular systolic dysfunction, and left ventricular diastolic dysfunction-each defined by specific inclusion and exclusion criteria. Participants will undergo a comprehensive microvascular assessment using investigational devices (including Perimed Periflux EPOS, PeriCam MultiFlow, and TCI P4) alongside stress cardiac magnetic resonance imaging (stress-CMR) for cardiac-specific evaluation.

DETAILED DESCRIPTION:
Non-invasive microvascular Assessment A comprehensive microvascular evaluation is performed using three investigational devices designed to capture detailed information on dermal perfusion. The Perimed Periflux 6000 EPOS employs diffuse reflectance spectroscopy (DRS) and laser Doppler flowmetry (LDF) for a single-point multi-modal assessment. The PeriCam MultiFlow performs imaging of dermal perfusion using multi-exposure laser contrast imaging (MELSCI) and measures blood oxygen saturation via multispectral imaging (MSI). Additionally, the TCI P4 utilizes spatial frequency domain imaging technology for quantification of perfusion and chromophore concentrations in the skin. Functional methods, including Post-Occlusive Reactive Hyperemia (PORH), Flow-Motion Analysis, and Thermal Provocation, are applied to assess dynamic microvascular responses.

Cardiac Magnetic Resonance Imaging (CMR) Stress#CMR is conducted using adenosine infusion and contrast enhancement to evaluate cardiac-specific microvascular function. This approach includes first-pass perfusion imaging and quantitative myocardial blood flow analyses, which allow for calculation of myocardial perfusion reserve.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the SCAPIS baseline (SCAPIS 1 study, 10 years ago)
* Cohort specific inclusion criteria apply, as stated in 'groups' section
* Has been invited to SCAPIS 2 core Singed informed consent to SCAPIS 2 core

Exclusion Criteria:

* Scarring, tattoos, or amputations that preclude device examination
* Cohort specific exclusion criteria apply, as stated in 'groups' section

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SCAPIS 2 General cohort
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Correlation between device-derived skin microcirculation variables and CCTA severity metrics including CAD-RADS (0-5) and plaque burden | Baseline
  Assess the correlation between skin microcirculation parameters measured by investigational devices (icluding PORH; 42°C local heat plateau; flow-motion endothelial-band power; iontophoresis acetylcholine response), coronary CT angiography (CCTA) severity metrics: CAD-RADS score, 0-5, zero is equivalent to no plaque and 5 indicates complete occlusionan (fully blocked) and Plaque burden indices (e.g., Segment Involvement Score [SIS])
  The device-derived microcirculation parameters are:
  Baseline perfusion, Perfusion after provocation, Peak perfusion, Time to peak, Recovery time, Capillary recruitment and Oxygen saturation (StO₂)
  The goal is to determine if these microcirculation measurements reflect coronary disease severity.
Discriminative performance of device-derived microcirculatory variables for significant coronary stenosis | Baseline
  Evaluate the ability of microcirculatory variables measured by investigational devices to discriminate between patients with and without significant coronary stenosis, defined as CAD-RADS ≥ 3 (≥50% luminal narrowing on coronary CT angiography).
Proportion of ANOCA participants (CAD-RADS <3 with angina per Rose questionnaire) who meet CMD criteria on stress-cardiac MRI using perfusion assessment | Baseline
  Calculate the proportion of participants classified as ANOCA (defined as CAD-RADS < 3 and angina symptoms per Rose Angina Questionnaire) who fulfill criteria for coronary microvascular dysfunction (CMD) based on stress cardiac MRI perfusion assessment according to site-standard protocols
Proportion of INOCA participants (CAD-RADS <3 with ishemia per Rose questionnaire) who meet CMD criteria on stress-cardiac MRI using perfusion assessment. | Baseline and at stress cardiac MRI- visit within 3 months
  Calculate the proportion of participants classified as INOCA (CAD-RADS < 3 and objective ischemia evidence) who fulfill CMD criteria based on stress cardiac MRI perfusion assessment..
Proportion of ANOCA participants who have INOCA | Baseline and at stress cardiac MRI- visit within 3 months
  Among participants identified with ANOCA (non-obstructive coronary artery disease on CT angiography), the proportion who demonstrate myocardial ischemia (INOCA) will be calculated. Ischemia will be assessed using cardiac MRI stress perfusion imaging, which is considered the gold standard for myocardial microcirculatory dysfunction
Assess whether peripheral microvascular function reflects myocardial perfusion abnormalities in CMD and mild CAD | Baseline and at stress cardiac MRI- visit within 3 months
  This outcome examines whether skin microcirculation parameters measured by investigational devices correlate with quantitative/ semiquantitative myocardial perfusion metrics obtained from stress cardiac-MRI in participants with:
  Coronary Microvascular Dysfunction (CMD) Non-obstructive coronary disease (CAD-RADS <3)
Correlation between investigational device variables and presence of Coronary Microvascular Dysfunction (CMD). | Baseline and at stress cardiac MRI- visit within 3 months
  Evaluate whether distinct cut-off values in device-derived microvascular parameters correlate with significant CMD. CMD will be defined by cardiac MRI stress perfusion imaging. The following variables will be assessed using investigational devices
Correlation of skin microcirculation variables with echocardiographic marker for diastolic function | Baseline
  Assess the general correlation between investigational device variables and E/é ratio (echocardiographic marker) to assess diastolic function.
  A high E/é ratio suggests elevated left atrial pressure and impaired relaxation (diastolic dysfunction).
  A low E/é ratio indicates normal filling pressures.
Association of skin microcirculation variables with elevated echocardiographic marker for diastolic dysfunction. | Baseline
  Determine whether investigationnal device-derived variables correlate with E/é > 15, indicative of increased left ventricular filling pressures.
Correlation of skin microcirculation variables with biomarker for cardiac stress | Baseline
  Assess general correlation between investigationnal device-derived variables and ProBNP as a biomarker of cardiac stress.
Association of skin microcirculation variables with elevated biomarker for measuring cardiac stress | Baseline
  Assess general correlation between investigationnal device-derived variables s and ProBNP as a biomarker of cardiac stress.
Identification of device variable thresholds predicting diastolic dysfunction/heart failure | Baseline and at stress cardiac MRI- visit within 3 months
  Evaluate whether specific cut-off values of investigational device-derived microcirculation variables are associated with confirmed dysfunction/heart failure
Correlation of skin microcirculation variables with high levels of a biomarker for average blood glucose | Baseline
  Calculate the correlation between the respective variables of the investigational devices and the incidence of HbA1c being > 65 mmol/mol.
Correlation of device-derived microcirculation variables with nephropathy | Baseline
  Calculate the correlation between the respective variables of the investigational devices and the incidence of nephropathy
Correlation betweed device-derived microcirculatory variables with endothelial/glycocalyx/inflammation biomarkers | Baseline
  Correlation between microcirculatory variables from investigational devices and biomarker panels (thrombomodulin, circulating endothelial cells, VE-cadherin, syndecan-1, hyaluronan, hsCRP, IL-6, GlycA).

SECONDARY OUTCOMES:
Correlation of Myogenic Response with Cardiovascular Disease | Baseline
  Asses the association between myogenic response from device-derived variables and cardiovascular disease incidence; includes incidence of myogenic vs endothelial dysfunction.
Association of Vascular Inflammation with Microcirculatory Variables | Baseline
  Correlation between systemic inflammation biomarkers (e.g., hsCRP, IL-6, GlycA) and device-derived microcirculatory measures; exploratory detection of early inflammatory alterations.
Mechanisms of endothelial damage and Cardiovascular Disease devlopment | Baseline
  Analysis of biomarker panels (endothelial/glycocalyx damage: thrombomodulin, VE-cadherin, syndecan-1, hyaluronan) to identify progression patterns and explore the correlation with device-derived microcirculatory variables.
Development of multi-modal Cardiovascular Disease risk score | Baseline
  Creation and validation of a composite risk score integrating microcirculatory variables derived from investigationa devices and biomarker data; evaluation of predictive performance for Cardiovascular Disease endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyd Hospital, Stockholm, Danderyd, Sweden

IPD SHARING:
Plan to Share IPD: Undecided